CLINICAL TRIAL: NCT06294587
Title: Evaluation of Free Gingival Graft Timing in Staged Guided Bone Regeneration: A Randomized Controlled Trial
Brief Title: Evaluation of Free Gingival Graft Timing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hussein Basma, Clinical Assistant Professor, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012407; UAB-SOD (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Ridge Augmentation; Alveolar Mucosa
Keywords: Ridge Augmentation; Attached mucosa; Dental implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FGG before GBR (Experimental): Free Gingival Graft(FGG) before the guided bone regeneration(GBR)
  Interventions: Procedure: FGG Before GBR
- FGG after GBR (Experimental): Free Gingival Graft(FGG) after the guided bone regeneration(GBR)
  Interventions: Procedure: FGG after GBR

INTERVENTIONS:
Procedure: FGG Before GBR — Free Gingival Graft before the guided bone regeneration,
  Arms: FGG before GBR
Procedure: FGG after GBR — Free Gingival Graft after the guided bone regeneration,
  Arms: FGG after GBR

SUMMARY:
This clinical trial aims to compare and evaluate the clinical outcomes between two distinct treatment sequences: free gingival graft surgery preceding guided bone regeneration and guided bone regeneration followed by free gingival graft.

DETAILED DESCRIPTION:
This clinical trial aims to compare and evaluate the clinical outcomes between two distinct treatment sequences: free gingival graft surgery preceding guided bone regeneration and guided bone regeneration followed by free gingival graft. The primary objective is to assess the influence of the tissue graft timing on the outcomes of the guided bone regeneration. The secondary goal is to compare the complications that may arise following the two procedures before implant placement.

ELIGIBILITY:
Inclusion Criteria:

* • At least 18 years old

  * No uncontrolled medical conditions or medications that will affect their bone healing.
  * Good oral hygiene is defined as a full-mouth plaque score ≤25%11.
  * Must be able to read and understand the informed consent document.
  * Has a need for implants to replace missing tooth/teeth in at least 1 quadrant of the mouth.
  * Insufficient alveolar ridge width for endosseous implant placement, defined as 5 mm or less, as determined by bone sounding and CBCT scan.
  * The patient and/or guardian is willing and able to comply with pre-operative and post-operative diagnostic and clinical evaluations required.
  * The patient is not pregnant or breastfeeding.

Exclusion Criteria:

* Active infectious diseases.

  * Liver or kidney dysfunction/failure.
  * Uncontrolled diabetes (HbA1c ≥ 8.5).
  * Active cancer treatment - such as active chemotherapy radiation therapy, or radiotherapy performed within ≤12 months from the procedure.
  * Taking medications that will affect their bone healing (for example, bisphosphonates and long-term anti-inflammatory medications).
  * Metabolic bone diseases that affect bone healing such as osteoporosis.
  * Pregnant or lactating women (self-reported).
  * Current tobacco and Marijuana smokers have 10 or more cigarettes per day, and former smokers (> 10 cigarettes) who quit < 10 ago (self-reported).
  * Poor oral hygiene.
  * Vertical loss of bone at the edentulous ridge.
  * History of periodontal disease.
  * The patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric outcome assessment | Baseline to 12 months
  The volumetric outcomes of interest will be volume change in mm3 (Vol) and the mean distance between the surface/mean thickness of the reconstructed volume in mm.
Buccal soft tissue profile | Baseline to 12 months
  The assessment involves measuring the profile of the buccal soft tissue from the implant shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States